CLINICAL TRIAL: NCT06518798
Title: Pilot Study on Fasting-Mimicking Diet in Asian Americans With Prediabetes
Brief Title: Feasibility and Preliminary Effects of Fasting-Mimicking Diet in Asian Americans With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Hannah Lui Park, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4223
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Prediabetes; Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fasting Mimicking Diet (FMD) (Experimental): The fasting-mimicking diet (FMD) group will be instructed on the benefits and use of the FMD kit. Participants will be given one 5-day FMD kit at their baseline visit. They will be instructed to follow the kit, and only eat its items, for five consecutive days and to report back for a follow-up visit and measurements at the end of their 5 days before returning to their normal diet.
  Interventions: Behavioral: Fasting Mimicking Diet

INTERVENTIONS:
Behavioral: Fasting Mimicking Diet — Participants will be instructed to follow their usual diet except for 5 days when they eat the foods in the FMD kit. The FMD consists of a blend of 100% plant based nutrients generally regarded as safe. One FMD kit provides for the replacement of the normal diet with plant products for five consecutive days. The formulation of these products was based on studies carried out at the Longevity Institute of the University of Southern California, led by Dr. Valter Longo and his collaborators over several decades of research.

SUMMARY:
This is a pilot study to determine the feasibility of studying the Fasting-Mimicking Diet (FMD), a dietary approach that involves the consumption of a specifically formulated, calorie-restricted nutrition regimen with a customized macronutrient composition, ratio, and quantity over a 5- day period, on a larger scale in Asian Americans with prediabetes and to examine the preliminary effects of the diet in study participants.

The main questions the study aims to answer are:

1. What are the recruitment, adherence, and attrition rates of eligible participants into the study?
2. Does one FMD cycle result in changes in fasting blood glucose levels and physical measurements in study participants?

Participants will be asked to undergo one cycle of FMD (for 5 days), fill out surveys, and come in for a pre-FMD and post-FMD study visit, during which physical measurements and fasting blood glucose and ketone levels will be measured.

ELIGIBILITY:
Inclusion criteria:

* Identify as Asian American
* Diagnosed with prediabetes according to at least one of the following:
* HbA1C 5.7%-6.4%
* Fasting blood glucose 100 to 125 mg/dL (5.6 to 6.9 mmol/L )
* Oral glucose tolerance test (OGTT) 140-199 mg/dL at two hours

Exclusion criteria:

* Individuals with a personal history of diabetes mellitus (ICD-10 codes E08-E13), cardiovascular disease, mental illness, drug dependency, pregnancy, and special dietary restrictions
* Individuals taking insulin or insulin-like drugs and individuals taking hypoglycemic agents other than metformin
* Individuals who are pregnant or breastfeeding
* Individuals with anaphylaxis food allergies
* Individuals who are allergic to tree nuts (macadamia, cashew, almond, pecan), soy, oats, sesame, or celery/celeriac
* Individuals who have completed the FMD in the past year

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | up to 6 months
  Recruitment rate will be determined based on the number of individuals who consented to be in the pilot Fasting Mimicking Diet trial per month.
Adherence rate | up to 6 months
  Study adherence will be assessed based on the participant's changes in fasting blood glucose and blood ketone levels measured pre- vs. post- Fasting Mimicking Diet (FMD); a post-FMD survey asking about adherence to the FMD; and attending the follow-up study appointment. The survey will also ask for participants' feedback on their experiences of the trial, including adverse events, and, if applicable, reasons for non-adherence, to enable further study optimization.
Attrition rate | up to 6 months
  Attrition rate will be determined based on the number of individuals who stopped consuming the Fasting Mimicking Diet or never started.
Willingness to participate in a future full Fasting Mimicking Diet (FMD) clinical trial | up to 6 months
  Willingness to participate in a future full FMD clinical trial (which would have 4 FMD cycles + additional study appointments at 4 months after the last FMD cycle) will also be assessed via survey at the conclusion of their participation in this pilot.

SECONDARY OUTCOMES:
Change in fasting blood glucose levels | Pre v. post 5-day FMD cycle
  Fasting blood glucose levels will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD) (using a lancet and glucose meter)
Change in blood pressure | Pre v. post 5-day FMD cycle
  Systolic and diastolic blood pressure will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD)
Change in body mass index | Pre v. post 5-day FMD cycle
  Body mass index will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD)
Change in percent body/visceral fat | Pre v. post 5-day FMD cycle
  Percent body fat and percent visceral fat will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD)
Change in waist circumference | Pre v. post 5-day FMD cycle
  Waist circumference will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD)
Change in ketone levels | Pre v. post 5-day FMD cycle
  β-Hydroxybutyrate level will be compared pre v. post 5 days of Fasting Mimicking Diet (FMD) using a lancet and blood ketone meter

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Lui Park, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Upon review by the study investigators

REFERENCES:
- [Background] Tabak AG, Herder C, Rathmann W, Brunner EJ, Kivimaki M. Prediabetes: a high-risk state for diabetes development. Lancet. 2012 Jun 16;379(9833):2279-90. doi: 10.1016/S0140-6736(12)60283-9. Epub 2012 Jun 9. PMID 22683128
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Sulaj A, Kopf S, von Rauchhaupt E, Kliemank E, Brune M, Kender Z, Bartl H, Cortizo FG, Klepac K, Han Z, Kumar V, Longo V, Teleman A, Okun JG, Morgenstern J, Fleming T, Szendroedi J, Herzig S, Nawroth PP. Six-Month Periodic Fasting in Patients With Type 2 Diabetes and Diabetic Nephropathy: A Proof-of-Concept Study. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2167-2181. doi: 10.1210/clinem/dgac197. PMID 35661214
- [Background] van den Burg EL, Schoonakker MP, van Peet PG, van den Akker-van Marle ME, Willems van Dijk K, Longo VD, Lamb HJ, Numans ME, Pijl H. Fasting in diabetes treatment (FIT) trial: study protocol for a randomised, controlled, assessor-blinded intervention trial on the effects of intermittent use of a fasting-mimicking diet in patients with type 2 diabetes. BMC Endocr Disord. 2020 Jun 24;20(1):94. doi: 10.1186/s12902-020-00576-7. PMID 32580710